CLINICAL TRIAL: NCT02243358
Title: A Neoadjuvant Phase II Study of Chemo-Radiotherapy in Patients With Resectable and Borderline Resectable Pancreatic Cancer
Brief Title: Phase II Study of Chemo-Radiotherapy in Patients With Resectable and Borderline Resectable Pancreatic Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Gazala Khan, MD, MD, Henry Ford Health System
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HFHS 13-03
Record Dates: First submitted 2014-09-04; First posted 2014-09-17 (Estimated); Results first posted 2023-10-27 (Actual); Last update posted 2023-10-27 (Actual); Status verified 2023-10

CONDITIONS: Pancreas Neoplasm Malignant Resectable
Keywords: Pancreatic, cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — Folfox protocol; 5-fluoropyrimidine; Gemcitabine; Radiotherapy; Pancreaticoduodenectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Neoadjuvant Chemo-Radiotherapy and Resection (Experimental): 2 cycles - FOLFOX6 (1 month) Gemcitabine/RT (5-6 weeks) Rest period 2 weeks Re-staging evaluation (CT scan to be done during the 2 weeks of rest) Surgery (To be performed no later than 6 weeks after completion of chemo-radiation)
  Interventions: Drug: Folfox6; Drug: Gemcitabine; Radiation: Radiation Therapy; Procedure: Pancreaticoduodenectomy with retroperitoneal lymphadenectomy

INTERVENTIONS:
Drug: Folfox6
  Other Names: 5 fluoropyrimidine
Drug: Gemcitabine
  Other Names: Gemzar
Radiation: Radiation Therapy
Procedure: Pancreaticoduodenectomy with retroperitoneal lymphadenectomy

SUMMARY:
To evaluate the safety and effectiveness of a novel neoadjuvant treatment strategy incorporating 5-fluorouracil/leucovorin with oxaliplatin ( FOLFOX )chemotherapy in combination with chemo-radiation with gemcitabine.

DETAILED DESCRIPTION:
The primary objective is to evaluate frequency of achieving complete resection ( RO resection )in patients with resectable and borderline resectable pancreatic cancer treated with a neoadjuvant regimen of FOLFOX followed by radiation therapy (RT) concurrent with gemcitabine chemotherapy at standard dosing.

Secondary objectives are to determine overall survival and progression-free survival as a function of time from study enrollment and to evaluate tolerability and toxicity of protocol treatment.

Eligible patients with resectable and borderline resectable pancreatic cancer will be accrued onto protocol therapy, which would include a neo-adjuvant phase followed by surgical resection. A cycle of FOLFOX treatment is 14 days. 2 cycles are intended prior to combined modality treatment. Combined modality treatment will begin 2 weeks (plus or minus 2 days) after the last FOLFOX administration. (Gemcitabine 1000mg/m² will be infused over 30 minutes on days 1, 8, 22, and 29 during the 5-week course of radiation treatment. The surgical procedure performed will be that required for a complete resection, and this will be based on the discretion of the operating surgeon. Patients will be followed for 1 year after completion of neoadjuvant therapy or until removal or termination from study, or until death, whichever occurs first. Patients will be seen in follow-up ever 3+/- 1 months for 1 year from completion of protocol therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically confirmed pancreatic adenocarcinoma of the pancreatic head or body
* Patients must have radiographically-confirmed surgically resectable or borderline resectable disease at study entry staged at T1-3, NO-1 and MO
* Age >/= 18years
* Life expectancy of greater than 6 months in the opinion of the investigator, excluding theh pancreatic cancer
* Eastern Cooperative Oncology Group (ECOG) performance status </= 1
* Required laboratory data (see protocol)
* Disease assessment by CT scan within 4 weeks of study entry
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Patients may not be receiving any other investigational agent
* Patients with metastatic disease are excluded from this clinical trial
* History of allergic reactions attributed to Fluorouracil (5FU), oxaliplatin and gemcitabine
* No prior chemotherapy or radiation therapy for pancreatic cancer (previous chemotherapy or radiation therapy for other malignancies is permitted)
* Patients with uncontrolled hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study.
* Uncontrolled serious intercurrent illness including, but not limited to, ongoing or serious active infection requiring IV antibiotics for over 30 days, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia other than chronic, stable atrial fibrillation, or psychiatric illness/social situations that would limit compliance with study requirements
* Pregnant or breastfeeding women are excluded from this study.
* Known HIV-positive patients are ineligible
* Patients with unresectable disease are excluded form the protocol (see Appendix B for National Comprehensive cancer Network [NCCN] criteria for determining resectability status). Surgical resectability must be confirmed by a surgeon experienced in pancreatic surgery.
* Patients with pancreatic tail lesions will be excluded

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2014-02; Primary Completion 2017-06-28 (Actual); Study Completion 2020-01-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gazala Khan, MD, Principal Investigator — Henry Ford Health System
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Through publication in peer reviewed journal

REFERENCES:
- [Result] Thanikachalam K, Damarla V, Seixas T, Dobrosotskaya I, Wollner I, Kwon D, Winters K, Raoufi M, Li J, Siddiqui F, Khan G. Neoadjuvant Phase II Trial of Chemoradiotherapy in Patients With Resectable and Borderline Resectable Pancreatic Cancer. Am J Clin Oncol. 2020 Jun;43(6):435-441. doi: 10.1097/COC.0000000000000688. PMID 32251119

RESULTS

PARTICIPANT FLOW:
Groups:
- Neoadjuvant Chemo-Radiotherapy and Resection: 2 cycles - FOLFOX6 (1 month) Gemcitabine/RT (5-6 weeks) Rest period 2 weeks Re-staging evaluation (CT scan to be done during the 2 weeks of rest) Surgery (To be performed no later than 6 weeks after completion of chemo-radiation)
  Folfox6
  Gemcitabine
  Radiation Therapy
  Pancreaticoduodenectomy with retroperitoneal lymphadenectomy
Period: Overall Study
Arm/Group | Neoadjuvant Chemo-Radiotherapy and Resection
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Neoadjuvant Chemo-Radiotherapy and Resection
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 64 [44 to 80]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 14
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race reported: White | 16
  Race reported: Black | 6
  Race reported: Hispanic | 1
  Race reported: Other | 1
Region of Enrollment [Number; unit: participants]
  United States | 24

OUTCOME MEASURES:

1. Primary Outcome: Frequency of R0 Resection
Description: Evaluate frequency of achieving R0 resection in patients with resectable and borderline resectable pancreatic cancer treated with a neoadjuvant regimen of FOLFOX followed by RT concurrent with gemcitabine chemotherapy at standard dosing
Time Frame: 6 weeks
Population: 13 patients underwent pancreatectomy after completion of neoadjuvant CRT
Measure: Count of Participants; unit: Participants
Arm/Group | Neoadjuvant Chemo-Radiotherapy and Resection
Number analyzed (Participants) | 13
Participants
  R0 resection | 11
  R1 resection | 2

ADVERSE EVENTS:
Time Frame: Consent to 1 year post completion of protocol therapy
Arm/Group | Neoadjuvant Chemo-Radiotherapy and Resection
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 21/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Neoadjuvant Chemo-Radiotherapy and Resection (N=24)
Anemia (Blood and lymphatic system disorders) | 2
Neutropenia (Blood and lymphatic system disorders) | 8
Thrombocytopenia (Blood and lymphatic system disorders) | 5
Fatigue (Metabolism and nutrition disorders) | 17
Nausea (Gastrointestinal disorders) | 21 (22)
Vomiting (Gastrointestinal disorders) | 9 (9)
Decreased appetite (Gastrointestinal disorders) | 10
Dehydration (Metabolism and nutrition disorders) | 4
Hypokalemia (Metabolism and nutrition disorders) | 4
Neuropathy (Nervous system disorders) | 6
Mucositis (Gastrointestinal disorders) | 3
Hypomagnesemia (Metabolism and nutrition disorders) | 2
Diarrhea (Gastrointestinal disorders) | 3
Cold intolerance (Nervous system disorders) | 2
Abdominal pain (Nervous system disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2013-03-11): https://cdn.clinicaltrials.gov/large-docs/58/NCT02243358/Prot_SAP_000.pdf